CLINICAL TRIAL: NCT05703373
Title: Increasing Access to Multiple Micronutrient Supplementation - A Pilot Intervention at up to 15 Clinics in Botswana
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ellen Caniglia, Assistant Professor of Epidemiology in Biostatistics and Epidemiology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 852412
Record Dates: First submitted 2022-12-22; First posted 2023-01-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple Micronutrient Supplement (MMS) supplied to clinic (Experimental)
  Interventions: Dietary Supplement: Multiple Micronutrient Supplement

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrient Supplement — Multiple micronutrient supplementation (MMS) which includes iron, folic acid, and additional micronutrients,

SUMMARY:
The purpose of this study is to pilot a clinic-level supplementation intervention at up to 15 antenatal clinics throughout Botswana. The overall objective of this study is to improve access to and uptake of MMS among pregnant women in Botswana. The investigators will evaluate both implementation outcomes (adoption, penetration, fidelity, and feasibility) and clinical outcomes (adverse birth outcomes, weight gain in pregnancy, and anemia) through linkage with the Tsepamo birth outcomes surveillance study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending interventional antenatal clinics during the 6-month study

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Proportion with first supplement filled by MMS | 6-month intervention period
  Among pregnant women presenting for their first antenatal visit during the 6-month intervention period at one of the intervention clinics who then deliver at one of the Tsepamo sites, the proportion for whom the first supplement filled during pregnancy is MMS. As comparators, we will use the 6-month pre-intervention period at the intervention clinics and the 6-month intervention period at non-intervention clinics (all non-intervention clinics as well as specific preselected control clinics).

SECONDARY OUTCOMES:
Implementation: Proportion for which MMS is filled | 6-month intervention period
  This outcome will be evaluated using data from clinic logbooks and by subtracting the number of supplements remaining in the clinic at the end of the study from the number of supplements provided to the clinic
Implementation: Proportion for which first and second supplement filled by MMS | 6-month intervention period
  Among pregnant women presenting for their first antenatal visit during the 6-month intervention period at one of the intervention clinics who then deliver at one of the Tsepamo sites, the proportion for whom MMS is filled at the first and second antenatal visit. This outcome will be evaluated through linkage with the Tsepamo Study. As comparators, we will use the 6-month pre-intervention period at the intervention clinics and the 6-month intervention period at non-intervention clinics (all non-intervention clinics as well as specific preselected control clinics).
Implementation: Feasibility | 8 months
  Feasibility of the intervention will be measured via qualitative pre- and post- intervention surveys among staff at the intervention clinics. Questions will be asked using a Likert scale ranging from completely disagree to completely agree. We will report the mean/median response for each question as well as the mean/median change in score between the pre and post surveys. As this is a qualitative measure there is no predefined minimum or maximum value.
Clinical: Number of Pregnant Women with an Adverse Birth Outcome | 6-months
  1) Any adverse birth outcome, consisting of stillbirth, preterm birth, SGA, neonatal death (as well as individual birth outcomes) among those who deliver at one of the Tsepamo sites. . As comparators, we will use the 6-month pre-intervention period at the intervention clinics and the 6-month intervention period at non-intervention clinics (all non-intervention clinics as well as specific preselected control clinics).
Clinical: Weight Gain in Pregnancy | 6-months
  Weight gain in pregnancy among those who deliver at one of the Tsepamo sites. As comparators, we will use the 6-month pre-intervention period at the intervention clinics and the 6-month intervention period at non-intervention clinics (all non-intervention clinics as well as specific preselected control clinics).
Clinical: Number of mothers diagnosed with Maternal Anemia | 6-months
  Number of mothers diagnosed with Anemia during the six month intervention or percentage of mothers diagnosed with anemia during 6 months of intervention compared to the percentage of mothers diagnosed with anemia in the 6 months prior to the intervention or 6 months after the interventions was completed.

CONTACTS AND LOCATIONS:
Locations (13):
- Botswana (13):
  - Kgatelopele (Block 8), Block 8, Gaborone
  - Gabarone West Clinic, Gaborone, Gaborone
  - Lesirane Clinic, Gaborone, Gaborone
  - Mahlaku Lekganyane (Mmopane Block 1), Gaborone, Gaborone
  - Nkoyaphiri Clinic, Gaborone, Gaborone
  - Tlokweng Main Clinic, Gaborone, Gaborone
  - Kopong Clinic, Kopong, Molepolole
  - Borakalalo, Molepolole, Molepolole
  - Boribamo Clinic, Molepolole, Molepolole
  - Boswelakoko-Borakalalo New Clinic, Molepolole, Molepolole
  - Phuthadikobo Clinic, Molepolole, Molepolole
  - Kediretswe Clinic, Palapye, Palapye
  - Palapye Primary Hospital, Palapye

IPD SHARING:
Plan to Share IPD: Undecided